CLINICAL TRIAL: NCT03012607
Title: Pharmacokinetics of Tenofovir in Blood, Plasma and Urine of Healthy Adults With Perfect, Median and Low Drug Adherence
Brief Title: Tenofovir Adherence to Rapidly Guide and Evaluate PrEP and HIV Therapy
Acronym: TARGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Chiang Mai University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Paul Drain, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000058; R21AI127200-01 (NIH)
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Hiv
Keywords: PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Perfect Adherence (Experimental): Participants will receive a single tablet of TENOFOVIR DISOPROXIL FUMARATE 300 Mg / EMTRICITABINE 200 Mg ORAL TABLET [TRUVADA] once daily for 6 weeks
  Interventions: Drug: Truvada
- Moderate Adherence (Experimental): Participants will receive a single tablet of TENOFOVIR DISOPROXIL FUMARATE 300 Mg / EMTRICITABINE 200 Mg ORAL TABLET [TRUVADA] 4 times per week (Monday, Wednesday, Friday, and Saturday) for 6 weeks
  Interventions: Drug: Truvada
- Poor Adherence (Experimental): Participants will receive a single tablet of TENOFOVIR DISOPROXIL FUMARATE 300 Mg / EMTRICITABINE 200 Mg ORAL TABLET [TRUVADA] 2 times per week (Monday, Thursday) for 6 weeks
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — Participants will be randomized into 1 of 3 groups (10 participants/group) to receive a controlled number of doses of tenofovir disoproxil fumarate (TDF, 300mg) in a combination pill with emtricitabine (FTC, 200mg) (Truvada®)

SUMMARY:
Adherence to antiretroviral therapy (ART) and pre-exposure prophylaxis (PrEP) are critical to the success of HIV treatment and therapeutic prevention. No accurate, objective point-of-care test is available to monitor adherence to either ART or PrEP. The inability to accurately identify poorly adherent patients will lead to more HIV infections (from failed PrEP and non-suppressive ART), more drug-resistant virus (selected by failing ART), and unnecessary switching to costly second- or third-line ART (when first-line regimens with virologic efficacy but non-adherence are stopped inappropriately). To address this critical knowledge gap, the investigators have developed a novel point-of-care test to detect the presence of tenofovir-the most common drug in both ART and PrEP treatments worldwide-in fingerprick blood or urine as an objective measure of ART and PrEP adherence.

Our central hypothesis is that the pharmacokinetics of tenofovir in blood and urine will support point-of-care tenofovir detection as an objective measure of adherence, and that our point-of-care tenofovir assay will have the ability to discriminate different drug adherence levels. The investigators will test our central hypotheses by pursuing the following two specific aims: (1) To assess our novel point-of-care tenofovir (TFV) assay in whole blood and urine specimens within a controlled pharmacokinetic study of HIV-negative adults receiving tenofovir disoproxil fumarate (TDF) with low, moderate, and perfect adherence; and (2) To validate our novel point-of-care tenofovir (TFV) assay on blood and urine specimens using an existing biorepository from a real-world clinical HIV prevention study.

This work is innovative because it develops an entirely new category of rapid diagnostic testing for monitoring ART and PrEP adherence at the clinical point of care. Our rapid assay will help clinicians identify patients in need of more adherence counseling, which when implemented will prevent HIV acquisition, emergence of drug resistant virus, and unnecessary ART regimen switching-measures that will improve national HIV programs and help preserve the global supply of an effective HIV medication.

DETAILED DESCRIPTION:
Objectives of the Study

Primary Objective:

• To determine the pharmacokinetics of tenofovir (TFV) in blood, urine and plasma in adults with perfect, median and low adherence to tenofovir disoproxil fumarate (TDF).

Secondary Objectives

* To determine the rate of tenofovir washout in blood, plasma and urine among participants with various levels of TDF adherence.
* To determine the steady-state concentrations of TFV in blood and plasma among controlled levels of TDF adherence.
* To compare the agreement between TFV in blood, plasma and urine concentrations.
* To determine the intracellular tenofovir-diphosphate (TFV-DP) trough concentrations in peripheral blood mononuclear cells (PBMC) and dried blood spot (DBS) samples in adults with perfect, median and low drug adherence.
* To identify possible concentration thresholds for the clinical interpretation of a binary point-of-care adherence test for measurement of TFV (and/or TFV-DP) in relation to adherence to TDF.

Design:

The study design is a randomized, open-label pharmacokinetic study in healthy adult volunteers. The study involves collection of clinical data and biological specimens, and subjects will provide written informed consent to participate. Healthy adult volunteers (HIV serology and hepatitis B surface Ag negative) will be enrolled. Once written consent is obtained, the screening visit will be performed. The study team will obtain each participant's phone number, address, and relevant contact information.

Screening Visit:

Participant screening will be performed within 14 days of enrollment. A detailed background demographic and health questionnaire will be administered. Ten mL of blood will be drawn for baseline assessments: complete blood count, HIV antibody testing, Hepatitis B surface Ag testing, renal and liver function tests and storage of blood in the biorepository. The blood and chemistry tests will be used to exclude subjects with any abnormal laboratory test among neutrophil count, hemoglobin, platelets, AST, or ALT. An abnormal test will be defined as Grade ≥3 by DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0 Nov. 2014). The results of the clinical examination and baseline laboratory assessments will be reviewed for inclusion/exclusion criteria.

Entry:

All entry visits will begin on a Monday morning. After receiving in-depth information on the study schedule, subjects meeting the inclusion criteria will be enrolled and randomized (1:1:1) into one of 3 groups to receive a controlled number of doses of Truvada® (Gilead Sciences Inc.), which contains tenofovir disoproxil fumarate (TDF, 300 mg) and emtricitabine (FTC, 200 mg) for 6 weeks. The participant will be carefully explained about their drug-dosing schedule, visit schedule and potential medication side effects.

We will enroll a total of 30 adults with evaluable PK samples (10 per group). All participants will start TDF in the morning of the Entry visit. The 6-week treatment period was chosen in order to ensure concentrations of tenofovir in the different matrices (i.e. blood, plasma, urine, PBMCs) mimic the expected conditions in patients with chronic dosing of perfect, median and low drug adherence. The blood/urine sampling schedule is based on the reported tenofovir plasma half-life and results of previous PK studies.

Tenofovir concentrations will be determined in each participant during three study phases (1) lead-in period, (2) intensive PK sampling, and (3) wash-out period.

Phase 1: Lead-in Period (Entry to 6 weeks) Visit Prior to 2nd Dose: Immediately prior to the second dose (i.e. Group 1: 24 post-dose (Day #2; Tuesday Morning); Group 2: 48 hours post-dose (Day #3; Wednesday Morning); and Group 3; 72 hours post-dose (Day #4; Thursday Morning) the subject will return to the hospital. A single blood sample will be drawn (5 mL). From this venous blood sample, 5 dried blood spots (50 µL/spot) will be prepared on a Whatman 903 filter paper card. The remaining blood will be centrifuged and the plasma stored. A single fingerstick whole blood sample will be collected and on a second Whatman 903 filter paper card 2 dried blood spots (50 µL/spot) will be prepared. A separate 10 mL blood drawn will be taken to collect PBMCs for determination of intracellular tenofovir-DP concentrations. Finally, a spot urine sample will be collected (5-10 mL). All samples will be stored at -70°C to -80°C.

Weeks 3 and 5 (both Monday morning, pre-dose): A single blood sample will be drawn (5 mL) prior to dose administration. From this venous blood sample, 5 dried blood spots (50 µL/spot) will be prepared on a Whatman 903 filter paper card. The remaining blood will be centrifuged and the plasma stored. A single fingerstick whole blood sample will be collected and 2 dried blood spots (50 µL/spot) will be prepared on a second Whatman 903 filter paper card. A separate 10 mL blood drawn will be taken to collect PBMCs for determination of intracellular tenofovir-DP concentrations. Finally, a spot urine sample will be collected (5-10 mL). All samples will be stored at -70°C to -80°C. Renal and liver function tests will be performed.

Phase 2: Intensive PK sampling (starting Monday morning of Week 7 for 24 hours) Week 7 Intensive PK visit: On the Monday morning of Week 7, subjects will return to the hospital in the early morning. A medical officer will conduct a physical examination and blood will be drawn for laboratory safety evaluations (AST, and ALT). Following their normal morning daily schedule of drug intake, a pre-dose blood sample will be drawn and a single Truvada® tablet will be administered on an empty stomach (at least 6 hour fast beforehand). This will be the last dose of Truvada® for all subjects. Venous blood (3 mL/time point) will be collected at 1, 2, 4, 6, 8, 10, 12, and 24 hours post-dose. At each time point, a venous blood DBS (5 spots) and fingerstick (2 spots) will be collected. Renal and liver function tests will be performed.

Urine samples will be collected pre-dose and over the intervals of 0-4 hours, 4-8 hours, 8-12 hours, and 12-24 hours. Subjects will have an additional 10 mL blood drawn pre-dose and PBMCs will be collected and stored at -70°C to -80°C. After 24 hours, the participant will be discharged from the hospital. The subject will be asked to collect all their urine until their next study visit in 24 hours.

Phase 3: Wash-out PK sampling (Weeks 7 to Week 10) Week 7 (Wednesday to Saturday): After the intensive PK sampling is complete, participants will return to the clinic once a day for the next 4 days (i.e. until the Saturday of Week 7) for a single venous blood draw (5mL), fingerprick sample collection for dried blood spot, and a spot urine sample (5-10 mL). The subject will be asked to collect all their urine until their next clinic visit.

Week 8 (Monday and Thursday): A single venous blood draw, fingerprick sample collection for dried blood spot, and a spot urine sample (5-10 mL) will be drawn on Monday and Thursday of Week 8. A single PBMC sample (10 mL blood) will be collected on Monday morning of week 8 (i.e. 1 week since last TDF dose).

Week 9 (Monday): A single venous blood draw, fingerprick sample collection for dried blood spot, and a spot urine sample (5-10 mL) will be drawn on Monday. A single PBMC sample (10 mL blood) will also be collected on Monday (i.e. 2 weeks since last TDF dose).

Week 10 (Monday): A single venous blood draw, fingerprick sample collection for dried blood spot, and a spot urine sample (5-10 mL) will be drawn on Monday. A single PBMC sample (10 mL blood) will also be collected on Monday morning (i.e. 3 weeks since last TDF dose).

End of Study visit (i.e. end of Week 10):

A single venous blood draw, fingerprick sample collection for dried blood spot, and a spot urine test (5-10 mL) will be drawn on Monday. A single PBMC sample (10 mL blood) will also be collected on Monday (i.e. 4 weeks since last TDF dose). A renal and liver function tests will be performed.

At this time the participants will have completed the study and no additional evaluations will be performed.

Tenofovir concentrations will be measured using validated liquid chromatography-triple quadrupole mass spectrometry (LC-MS/MS) assays at the Faculty of Associated Medical Sciences at Chiang Mai University. Intracellular tenofovir-diphosphate (TFV-DP) concentrations will be determined using a validated a LC-MS based assay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and <50 years old
* HIV and Hepatitis B surface Ag negative
* Normal renal function (estimated GFR >60 mL/min by the Cockcroft-Gault equation)
* Willing/able to provided written informed consent

Exclusion Criteria:

* Pregnant female
* Any significant lab abnormality of neutrophil count, hemoglobin, platelets, AST, or ALT (Defined as Grade ≥3 by DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0, Nov. 2014)
* History of using PrEP or thought to be eligible to receive PrEP.
* Any clinically significant diseases or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, might compromise participation in this study
* Any concurrent participation in another clinical trial

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Truvada concentration | 24, 48, 72 hours post-dose
  Area under the plasma concentration versus time curve (AUC) of Truvada concentration

SECONDARY OUTCOMES:
Maximum plasma concentration of Truvada | 24, 48, 72 hours post-dose
  Maximum plasma concentration of Truvada
Renal clearance of Truvada | 24, 48, 72 hours post-dose
  Renal clearance of Truvada
Time to Maximum Plasma Concentration(Cmax) of Truvada | 24, 48, 72 hours post-dose
  Time to Maximum Plasma Concentration(Cmax) of Truvada

CONTACTS AND LOCATIONS:
Overall Officials: Paul Drain, MD, MPH, Principal Investigator — University of Washington; Tim R Cressey, PhD, Principal Investigator — Chiang Mai University; Oraphan Siriprakaisil, MD, Principal Investigator — Sanpatong Hospital, Chiang Mai; Virat Klinbuayaem, MD, Principal Investigator — Sanpatong Hospital, Chiang Mai
Locations (1):
- Sanpatong Hospital, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
We will make decisions to share IPD on case by case basis

REFERENCES:
- [Derived] Drain PK, Kubiak RW, Siriprakaisil O, Klinbuayaem V, Quame-Amaglo J, Sukrakanchana PO, Tanasri S, Punyati P, Sirirungsi W, Cressey R, Bacchetti P, Okochi H, Baeten JM, Gandhi M, Cressey TR. Urine Tenofovir Concentrations Correlate With Plasma and Relate to Tenofovir Disoproxil Fumarate Adherence: A Randomized, Directly Observed Pharmacokinetic Trial (TARGET Study). Clin Infect Dis. 2020 May 6;70(10):2143-2151. doi: 10.1093/cid/ciz645. PMID 31314073
- [Derived] Cressey TR, Siriprakaisil O, Klinbuayaem V, Quame-Amaglo J, Kubiak RW, Sukrakanchana PO, Than-In-At K, Baeten J, Sirirungsi W, Cressey R, Drain PK. A randomized clinical pharmacokinetic trial of Tenofovir in blood, plasma and urine in adults with perfect, moderate and low PrEP adherence: the TARGET study. BMC Infect Dis. 2017 Jul 14;17(1):496. doi: 10.1186/s12879-017-2593-4. PMID 28705153